CLINICAL TRIAL: NCT05604001
Title: In-office Hysteroscopic Laser Ablation for Symptomatic Submucous Uterine Fibroids: Impact on Size and Vascularization.
Brief Title: In-office Hysteroscopic Laser Ablation for Symptomatic Submucous Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Responsible Party: Principal Investigator, Sergio Haimovich, Director of the Gynecology Department at the Laniado Hospital, Ariel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LaMyA
Record Dates: First submitted 2022-10-23; First posted 2022-11-03 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Laser Hysteroscopic Ablation of Submucous Myoma

STUDY DESIGN:
Intervention Model Description: patients with symptomatic submucosal fibroides were elected for hysteroscopy laser ablation of the fibroid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptomatic submucosal myoma (Experimental): patients with symptomatic submucosal fibroids (heavy menstrual bleeding) were elected for hysteroscopy with laser ablation of the myoma.
  Interventions: Device: hysteroscopic ablation of submucous uterine fibroid using diode laser

INTERVENTIONS:
Device: hysteroscopic ablation of submucous uterine fibroid using diode laser — patients with symptomatic submucosal fibroids (heavy menstrual bleeding) were elected for hysteroscopy and laser ablation of the myoma

SUMMARY:
To evaluate feasibility and efficacy of in-office hysteroscopic ablation of submucous uterine fibroid using diode laser

DETAILED DESCRIPTION:
A pilot study was conducted between January 2018 and January 2019 in a tertiary care university hospital. Patients with at least one symptomatic, class 0-2 of FIGO classification, uterine fibroid of ≤ 7cm in size were eligible for inclusion. Evaluation of the changes in fibroid size and vascularity was performed using 3D Doppler ultrasonography. Vaporization of the fibroid core was conducted using a 1470nm wavelength diode laser inserted through the hysteroscope's working channel. Primary outcome was the evaluation of the fibroid volume before and at 2 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients without desire of future fertility (symptoms included heavy menstrual bleeding, abdominal discomfort, bulk symptoms such as urinary frequency, pelvic pressure and constipation),
* grade 0-2 (FIGO classification) ≤ 7cm fibroids with evident vascularity seen by 3D-DS compared to its adjacent myometrial tissue

Exclusion Criteria:

* intramural fibroids (FIGO class 3 or more),
* >2 submucosal fibroids,
* pelvic inflammatory disease,
* known gynecologic malignancy,
* severe cervical stenosis,
* pregnancy
* desire of future fertility,
* previous cervical surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — fiborid is a pathology that affects women´s uterus
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Bleeding | before the procedure and at 3 months follow up visit
  improvement of the heavy menstrual bleeding

SECONDARY OUTCOMES:
fibroid volume reduction | before the procedure and at 3 months follow up visit
  measure by US the reduction of the myoma size
changes on the myoma vascularity | before the procedure and at 3 months follow up visit
  measure by 3D US Doppler Color

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Haimovich, MD, PhD, Principal Investigator — Laniado University Hospital - Ariel University
Locations (4):
- Laniado University Hospital, Netanya, Israel
- Italy (2):
  - University of Cagliari, Cagliari
  - universita della campagna luigi Vanvitelli, Napoli
- Parc de Salut Mar, Barcelona, Spain

REFERENCES:
- [Background] Carranza-Mamane B, Havelock J, Hemmings R; REPRODUCTIVE ENDOCRINOLOGY AND INFERTILITY COMMITTEE; SPECIAL CONTRIBUTOR. The management of uterine fibroids in women with otherwise unexplained infertility. J Obstet Gynaecol Can. 2015 Mar;37(3):277-285. doi: 10.1016/S1701-2163(15)30318-2. PMID 26001875
- [Background] Valentine LN, Bradley LD. Hysteroscopy for Abnormal Uterine Bleeding and Fibroids. Clin Obstet Gynecol. 2017 Jun;60(2):231-244. doi: 10.1097/GRF.0000000000000287. PMID 28406809
- [Background] Capmas P, Levaillant JM, Fernandez H. Surgical techniques and outcome in the management of submucous fibroids. Curr Opin Obstet Gynecol. 2013 Aug;25(4):332-8. doi: 10.1097/GCO.0b013e3283630e10. PMID 23812380
- [Background] Yendru KS, Yelamanchi SD, Vaddiraju GB. Hysteroscopic Resection of Submucous Fibroids in Symptomatic Women. J Obstet Gynaecol India. 2019 Apr;69(2):166-172. doi: 10.1007/s13224-018-1139-z. Epub 2018 May 31. PMID 30956472
- [Background] Vitale SG, Lagana AS, Caruso S, Garzon S, Vecchio GM, La Rosa VL, Casarin J, Ghezzi F. Comparison of three biopsy forceps for hysteroscopic endometrial biopsy in postmenopausal patients (HYGREB-1): A multicenter, single-blind randomized clinical trial. Int J Gynaecol Obstet. 2021 Dec;155(3):425-432. doi: 10.1002/ijgo.13669. Epub 2021 Apr 4. PMID 33686708
- [Background] Nappi L, Pontis A, Sorrentino F, Greco P, Angioni S. Hysteroscopic metroplasty for the septate uterus with diode laser: a pilot study. Eur J Obstet Gynecol Reprod Biol. 2016 Nov;206:32-35. doi: 10.1016/j.ejogrb.2016.08.035. Epub 2016 Aug 31. PMID 27632410
- [Background] Haimovich S, Lopez-Yarto M, Urresta Avila J, Saavedra Tascon A, Hernandez JL, Carreras Collado R. Office Hysteroscopic Laser Enucleation of Submucous Myomas without Mass Extraction: A Case Series Study. Biomed Res Int. 2015;2015:905204. doi: 10.1155/2015/905204. Epub 2015 May 18. PMID 26090457
- [Background] Goldfarb HA. Laparoscopic coagulation of myoma (myolysis). Obstet Gynecol Clin North Am. 1995 Dec;22(4):807-19. No abstract available. PMID 8786884
- [Background] Donnez J, Squifflet J, Polet R, Nisolle M. Laparoscopic myolysis. Hum Reprod Update. 2000 Nov-Dec;6(6):609-13. doi: 10.1093/humupd/6.6.609. PMID 11129695
- [Background] Dubuisson JB, Chapron C, Fauconnier A, Kreiker G. Laparoscopic myomectomy and myolysis. Curr Opin Obstet Gynecol. 1997 Aug;9(4):233-8. PMID 9263713
- [Background] D'Alterio MN, Scicchitano F, Fanni D, Faa G, Laganà AS, Noventa M, et al. Ex vivo myolysis with dual wavelengths diode laser system: macroscopic and histopathological examination. CEOG. 2021;48(4):875-82
- [Background] Nieuwenhuis LL, Hehenkamp WJK, Brolmann HAM, Huirne JAF. 3D power Doppler in uterine fibroids; influence of gain, cardiac cycle and off-line measurement techniques. J Obstet Gynaecol. 2018 Jan;38(1):103-109. doi: 10.1080/01443615.2017.1330323. Epub 2017 Aug 7. PMID 28780884
- [Background] Vitale SG, Lagana AS, Torok P, Lasmar RB, Carugno J, Palumbo M, Tesarik J. Virtual sonographic hysteroscopy in assisted reproduction: A retrospective cost-effectiveness analysis. Int J Gynaecol Obstet. 2022 Jan;156(1):112-118. doi: 10.1002/ijgo.13651. Epub 2021 Mar 16. PMID 33615469
- [Background] Fleischer AC. Sonographic depiction of tumor vascularity and flow: from in vivo models to clinical applications. J Ultrasound Med. 2000 Jan;19(1):55-61. doi: 10.7863/jum.2000.19.1.55. PMID 10625191
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Background] Munro MG, Critchley HO, Broder MS, Fraser IS; FIGO Working Group on Menstrual Disorders. FIGO classification system (PALM-COEIN) for causes of abnormal uterine bleeding in nongravid women of reproductive age. Int J Gynaecol Obstet. 2011 Apr;113(1):3-13. doi: 10.1016/j.ijgo.2010.11.011. Epub 2011 Feb 22. PMID 21345435
- [Background] Carugno J, Grimbizis G, Franchini M, Alonso L, Bradley L, Campo R, Catena U, Carlo A, Attilio DSS, Martin F, Haimovich S, Isaacson K, Moawad N, Saridogan E, Clark TJ. International Consensus Statement for Recommended Terminology Describing Hysteroscopic Procedures. J Minim Invasive Gynecol. 2022 Mar;29(3):385-391. doi: 10.1016/j.jmig.2021.10.004. Epub 2021 Oct 12. PMID 34648932
- [Background] Bettocchi S, Selvaggi L. A vaginoscopic approach to reduce the pain of office hysteroscopy. J Am Assoc Gynecol Laparosc. 1997 Feb;4(2):255-8. doi: 10.1016/s1074-3804(97)80019-9. PMID 9050737
- [Background] Tinelli R, Litta P, Angioni S, Bettocchi S, Fusco A, Leo L, Landi S, Cicinelli E. A multicenter study comparing surgical outcomes and ultrasonographic evaluation of scarring after laparoscopic myomectomy with conventional versus barbed sutures. Int J Gynaecol Obstet. 2016 Jul;134(1):18-21. doi: 10.1016/j.ijgo.2015.10.029. Epub 2016 Mar 31. PMID 27209335
- [Background] Vitale SG, Riemma G, Haimovich S, Carugno J, Alonso Pacheco L, Perez-Medina T, Parry JP, Torok P, Tesarik J, Della Corte L, Cobellis L, Di Spiezio Sardo A, De Franciscis P. Risk of endometrial cancer in asymptomatic postmenopausal women in relation to ultrasonographic endometrial thickness: systematic review and diagnostic test accuracy meta-analysis. Am J Obstet Gynecol. 2023 Jan;228(1):22-35.e2. doi: 10.1016/j.ajog.2022.07.043. Epub 2022 Aug 4. PMID 35932873
- [Background] Georgiou D, Tranoulis A, Jackson TL. Hysteroscopic tissue removal system (MyoSure) for the resection of polyps, sub-mucosal leiomyomas and retained products of conception in an out-patient setting: A single UK institution experience. Eur J Obstet Gynecol Reprod Biol. 2018 Dec;231:147-151. doi: 10.1016/j.ejogrb.2018.10.030. Epub 2018 Oct 12. PMID 30388609
- [Background] Munro MG. Uterine polyps, adenomyosis, leiomyomas, and endometrial receptivity. Fertil Steril. 2019 Apr;111(4):629-640. doi: 10.1016/j.fertnstert.2019.02.008. PMID 30929720
- [Background] Vilos GA, Vilos AG, Abu-Rafea B, Leyland N, Allaire C, Laberge PY, Murji A, Singh SS, Thiel J. Interventional Uterine-Sparing Therapies for Leiomyomas: A Commentary on Myolysis. J Obstet Gynaecol Can. 2020 Feb;42(2):169-172. doi: 10.1016/j.jogc.2019.08.025. Epub 2019 Nov 23. PMID 31767379